CLINICAL TRIAL: NCT00946153
Title: Phase I/II Study of E7080 in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Study of Lenvatinib (E7080) in Participants With Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-202
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma; Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma | interventions — lenvatinib

ARMS (1):
- Lenvatinib (Experimental)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — In the Dose-Escalation Component of the study, lenvatinib will be administered as continuous once-daily oral dosing. Dose-escalation will occur based on safety information obtained during Cycle 1. The recommended dose for the Expansion Component of the study will use the MTD in Cycle 1.
  Other Names: E7080

SUMMARY:
The purpose of this study is to determine maximum tolerated dose (MTD), efficacy, safety and tolerability, pharmacokinetics, pharmacodynamics, and anti-tumor effect of E7080 when is administered continually once daily in participants with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or clinically confirmed diagnosis of advanced HCC.
2. Eastern Cooperative Oncology Group-Performance Status (ECOG-PS): 0-1.
3. Adequate laboratory values/organ function tests.

Exclusion criteria:

1. Simultaneous or metachronous cancers.
2. Pericardial, ascites, or pleural effusion requiring drainage.
3. Brain metastasis/meningeal carcinomatosis presenting clinical symptoms or requiring treatment.
4. Malabsorption syndrome.
5. Artery-portal vein shunt or artery-vein shunt preventing proper diagnosis of tumor.
6. Use of drugs known to inhibit cytochrome P3A4.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-07-24 (Actual); Primary Completion 2014-06-15 (Actual); Study Completion 2015-08-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (10):
  - Kashiwa-shi, Chiba
  - Kurume-shi, Fukuoka
  - Sapporo, Hokkaido
  - Kawasaki-shi, Kanagawa
  - Osaka, Osaka
  - Osakasayama-shi, Osaka
  - Saga, Saga-ken
  - Chuo-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino-shi, Tokyo
- South Korea (2):
  - Gangnam-gu, Seoul
  - Songpa-gu, Seoul

REFERENCES:
- [Derived] Ikeda K, Kudo M, Kawazoe S, Osaki Y, Ikeda M, Okusaka T, Tamai T, Suzuki T, Hisai T, Hayato S, Okita K, Kumada H. Phase 2 study of lenvatinib in patients with advanced hepatocellular carcinoma. J Gastroenterol. 2017 Apr;52(4):512-519. doi: 10.1007/s00535-016-1263-4. Epub 2016 Oct 4. PMID 27704266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 sites in Japan and 2 sites in South Korea from 24 Jul 2009 to 13 Aug 2015.
Groups:
- Phase 1: Group 1: Lenvatinib: 12 mg: Participants with child-pugh (CP) scores of 5 or 6 received a starting dose of 12 milligram (mg) (three 4 mg tablets) lenvatinib orally once daily (QD) in a 28-day treatment cycle in the dose-escalation scheme (group 1) on an empty stomach or at least 1 hour after eating until the tolerated dose was achieved.
- Phase 1: Group 1: Lenvatinib: 16 mg: Participants with CP scores of 5 or 6 received 16 mg (four 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-escalation scheme (group 1) on an empty stomach or at least 1 hour after eating.
- Phase 1: Group 2: Lenvatinib: 8 mg: Participants with CP scores of 7 or 8 received 8 mg (two 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle which was the lowest dose at which tolerability was confirmed in group 1, was used as the starting dose in the dose-determination scheme (group 2) on an empty stomach or at least 1 hour after eating.
- Phase 1: Group 2: Lenvatinib: 12 mg: Participants with CP scores of 7 or 8 received 12 mg (three 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-determination scheme (group 2) on an empty stomach or at least 1 hour after eating.
- Phase 2: Lenvatinib: 12 mg: Participants with CP scores of 5 or 6 received recommended dose (RD) of 12 mg (three 4 mg tablets) lenvatinib established from group 1, in the dose escalation component (phase 1) study, orally QD in a 28-day treatment cycle in dose expansion component on an empty stomach or at least 1 hour after eating.
Period: Phase 1
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group 1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg | Phase 2: Lenvatinib: 12 mg
Started | 6 | 3 | 6 | 5 | 0
Completed | 6 | 3 | 6 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group 1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg | Phase 2: Lenvatinib: 12 mg
Started | 0 | 0 | 0 | 0 | 46
Completed | 0 | 0 | 0 | 0 | 33
Not Completed | 0 | 0 | 0 | 0 | 13
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 6
Not completed — Need more reduction of dose | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — 14 days washout for recovery due to AE | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of lenvatinib, and had at least 1 post baseline efficacy evaluation.
Groups:
- Phase 1: Group 1: Lenvatinib: 12 mg: Participants with CP scores of 5 or 6 received a starting dose of 12 mg (three 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-escalation scheme (group 1) on an empty stomach or at least 1 hour after eating until the tolerated dose was achieved.
- Phase 2: Lenvatinib: 12 mg: Participants with CP scores of 5 or 6 received RD of 12 mg (three 4 mg tablets) lenvatinib established from group 1, in the dose escalation component (phase 1) study, orally QD in a 28-day treatment cycle in dose expansion component on an empty stomach or at least 1 hour after eating.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group 1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg | Phase 2: Lenvatinib: 12 mg | Total
Number analyzed (Participants) | 6 | 3 | 6 | 5 | 46 | 66
Age, Customized [Count of Participants; unit: Participants]
  >=37 years and <=80 years | 6 | 3 | 6 | 5 | 46 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 13 | 16
  Male | 5 | 1 | 6 | 5 | 33 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 6 | 5 | 46 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Lenvatinib
Description: The MTD was defined as the highest dose level at which no more than 1 of 6 participants had a dose limiting toxicities (DLT). DLT was defined as any of the following events: grade 4 or higher hematologic toxicity or grade 3 thrombocytopenia that required blood transfusion, grade 3 or higher nonhematologic toxicity, grade 4 hypertension uncontrolled by antihypertensive drug(s), aspartate aminotransferase/alanine aminotransferase (AST/ALT) greater than (>) 10.0*upper limit of normal (ULN), proteinuria 4+ by urine dipstick, proteinuria 3+ by urine dipstick was to be monitored by 24-hour urine collection, proteinuria >3.5 gram (g) for 24 hours, diarrhea/vomiting/nausea of grade 3 or higher that was uncontrollable despite maximal supportive therapies and abnormal clinical laboratory values that required no treatment, grade 3 proteinuria by dipstick, diarrhea/vomiting/nausea that was managed with supportive therapies were not considered as DLT.
Time Frame: Up to 28 days (Cycle1)
Population: Safety analysis set (SAS) included all participants who received at least 1 dose of lenvatinib, and had at least 1 post baseline safety evaluation.
Measure: Number; unit: milligram (mg)
Groups:
- Phase 1: Group 1: Levatinib 12 or 16 mg (CP Score 5 or 6): Participants with CP scores of 5 or 6 received 12 mg (three 4 mg tablets) or 16 mg (four 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-escalation scheme (group 1) on an empty stomach or at least 1 hour after eating.
- Phase 1: Group 2: Lenvatinib 8 or 12 mg (CP Score 7 or 8): Participants with CP scores of 7 or 8 received 8 mg (two 4 mg tablets) or 12 mg (three 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-determination scheme (group 2) on an empty stomach or at least 1 hour after eating.
Arm/Group | Phase 1: Group 1: Levatinib 12 or 16 mg (CP Score 5 or 6) | Phase 1: Group 2: Lenvatinib 8 or 12 mg (CP Score 7 or 8)
Number analyzed (Participants) | 9 | 11
milligram (mg) | 12 | 8

2. Primary Outcome: Phase 2: Time to Progression (TTP) by Independent Review Assessment
Description: TTP was defined as the time from the date of registration to the date when progressive disease (PD) was first confirmed. PD was evaluated according to modified response evaluation criteria in solid tumors (mRECIST) by an independent imaging review. PD was defined as at least a 20 percent (%) increase in the sum of long diameter (LD) of target lesions as compared with the smallest sum of LD and the increase of LD was at least 5 millimeter (mm) (including new lesions).
Time Frame: From day of registration to the day when PD was first confirmed (approximately up to 6.1 years)
Population: Per protocol set (PPS) included all participants in full analysis set (FAS), who showed greater than or equal to (>=) 75% cumulative treatment compliance, had a baseline and post baseline tumor response assessment, and completed at least 2 cycles or discontinued during the 2 cycles due to PD or death.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2 : Lenvatinib :12 mg: Participants with CP scores of 5 or 6 received lenvatinib RD of 12 mg (three 4 mg tablets) established from group 1 in the dose escalation component (Phase 1) study, orally QD in a 28-day treatment cycle in dose expansion component on an empty stomach or at least 1 hour after eating.
Arm/Group | Phase 2 : Lenvatinib :12 mg
Number analyzed (Participants) | 41
months | 7.40 [5.50 to 9.40]

3. Secondary Outcome: Phase 1: Best Overall Response (BOR) of Lenvatinib by Investigator Assessment
Description: BOR was performed using RECIST1.1 and was measured as complete response (CR) defined as when an overall response of CR was obtained 2 or more consecutive times at intervals of at least 28 days (the date when the second overall response of CR was confirmed and the BOR established as CR was regarded as the "CR confirmed date), partial response (PR) defined as when the overall response of PR or better (CR or PR) was obtained 2 or more consecutive times at intervals of at least 28 days (the date when the second overall response of PR was confirmed and the BOR established as PR will be regarded as the "PR confirmed date), PD defined as when the BOR was neither CR, PR, or stable disease (SD), and the overall response was PD, SD defined as when the BOR obtained was neither CR nor PR, but no PD from the initial administration to the end of Cycle 2 and the overall response of SD or better occurred at least once and not evaluable (NE) was when the overall response was NE in all cases.
Time Frame: Every 8 weeks (approximately up to 18.4 months)
Population: Efficacy analysis set (EAS) included all participants who received at least 1 dose of lenvatinib, and had at least 1 postbaseline efficacy evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Group1: Lenvatinib: 16 mg: Participants with CP scores of 5 or 6 received 16 mg (four 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-escalation scheme (group 1) on an empty stomach or at least 1 hour after eating.
- Phase 1: Group 2: Lenvatinib: 8 mg: Participants with CP scores of 7 or 8 received 8 mg (two 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle which was the lowest dose at which tolerability was confirmed in group1, was used as the starting dose in the dose-determination scheme (group 2) on an empty stomach or at least 1 hour after eating.
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg
Number analyzed (Participants) | 6 | 3 | 6 | 5
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 1 | 1 | 0
  Stable Disease | 2 | 2 | 4 | 2
  Progressive Disease | 2 | 0 | 1 | 3
  Not Evaluable | 1 | 0 | 0 | 0

4. Secondary Outcome: Phase 1: Objective Response Rate (ORR) by Investigator Assessment
Description: ORR was defined as the percentage of participants who achieved a tumor response measured by RECIST 1.1 of CR defined as disappearance of all target lesions (a short diameter is less than (<)10 mm if it exists in a lymph node) plus PR defined as at least 30% decrease in the sum of the long diameter LD (hereafter referred to as sum of LD) of all target lesions, as compared with Baseline summed LD.
Time Frame: From day of registration to the day when PD was first confirmed or death (approximately 6.1 years)
Population: EAS included participants who received at least 1 dose of lenvatinib, and had at least 1 postbaseline efficacy evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg
Number analyzed (Participants) | 6 | 3 | 6 | 5
percentage of participants | 16.7 | 33.3 | 16.7 | 0

5. Secondary Outcome: Phase 1: Disease Control Rate (DCR) by Investigator Assessment
Description: DCR was measured by RECIST 1.1 and defined as CR which was defined as disappearance of all target lesions (a short diameter was <10 mm if it exists in a lymph node) plus PR which was defined as at least 30% decrease in the sum of the long diameter (hereafter referred to as sum of LD) of all target lesions, as compared with baseline summed LD plus SD which was reduction in tumor volume of less than 50% or an increase in the volume of 1 or more measurable lesions of less than 25% without the appearance of any new lesions which was neither tumor shrinkage corresponding to PR nor tumor expansion corresponding to PD.
Time Frame: Up to Week 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg
Number analyzed (Participants) | 6 | 3 | 6 | 5
percentage of participants | 50 | 100 | 83.3 | 40.0

6. Secondary Outcome: Phase 2: Progression-free Survival (PFS) by Independent Review Assessment
Description: PFS was defined as the time from the date of registration until the date when PD was first confirmed or death (whichever occurred first) as determined by mRECIST and PD was defined as at least a 20% increase in the sum of long diameters of target lesions, taking as reference the baseline sum of diameters of target lesions.
Time Frame: From day of registration to the day when PD was first confirmed or death (approximately 6.1 years)
Population: PPS included all participants in the FAS who showed >=75% cumulative treatment compliance, had a baseline and post baseline tumor response assessment, and completed at least 2 cycles or discontinued during the 2 cycles due to PD or death.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2 : Lenvatinib :12 mg: Participants with CP scores of 5 or 6 received RD of 12 mg (three 4 mg tablets) lenvatinib established from group 1 in the dose escalation component (phase 1) study, orally QD in a 28-day treatment cycle in dose expansion component on an empty stomach or at least 1 hour after eating.
Arm/Group | Phase 2 : Lenvatinib :12 mg
Number analyzed (Participants) | 41
months | 7.40 [5.50 to 9.40]

7. Secondary Outcome: Phase 2: Objective Response Rate (ORR) by Independent Review Assessment
Description: ORR was defined as the percentage of participants who achieved a tumor response measured by mRECIST of CR defined as disappearance of all target lesions (a short diameter is <10 mm if it exists in a lymph node) plus PR defined as at least 30% decrease in the sum of the long diameter LD (hereafter referred to as sum of LD) of all target lesions, as compared with Baseline summed LD.
Time Frame: From day of registration to the day when PD was first confirmed or death (approximately 6.1 years)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 : Lenvatinib :12 mg
Number analyzed (Participants) | 41
percentage of participants | 41.5 [26.3 to 57.9]

8. Secondary Outcome: Phase 2: Disease Control Rate (DCR) by Independent Review Assessment
Description: DCR was measured by mRECIST and defined as CR which was defined as disappearance of all target lesions (a short diameter is <10 mm if it exists in a lymph node) plus PR which was defined as at least 30% decrease in the sum of the long diameter (hereafter referred to as sum of LD) of all target lesions, as compared with baseline summed LD plus SD which was reduction in tumor volume of less than 50% or an increase in the volume of 1 or more measurable lesions of less than 25% without the appearance of any new lesions which was neither tumor shrinkage corresponding to PR nor tumor expansion corresponding to PD.
Time Frame: Weeks 8 and 16
Population: PPS included all participants in the FAS showed >=75% cumulative treatment compliance, had a baseline and post baseline tumor response assessment, and completed at least 2 cycles or discontinued during the 2 cycles due to PD or death.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Phase 2 : Lenvatinib :12 mg
Number analyzed (Participants) | 41
percentage of participant
  Week 8 | 87.8 [73.8 to 95.9]
  Week 16 | 78.0 [62.4 to 89.4]

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of registration until the date of death.
Time Frame: From day of registration to the day of death (approximately 6.1 years)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 : Lenvatinib :12 mg
Number analyzed (Participants) | 41
months | 18.30 [12.70 to 25.10]

ADVERSE EVENTS:
Time Frame: From start of study drug administration until approximately up to 6.1 years
Groups:
- Phase 1: Group 1: Lenvatinib: 12 mg: Participants with child CP scores of 5 or 6 received a starting dose of 12 mg (three 4 mg tablets) lenvatinib orally QD in a 28-day treatment cycle in the dose-escalation scheme (group 1) on an empty stomach or at least 1 hour after eating until the tolerated dose was achieved.
- Phase 2: Lenvatinib: 12 mg: Participants with CP scores of 5 or 6 received lenvatinib RD of 12 mg (three 4 mg tablets) established from group 1 in the dose escalation component (Phase1) study, orally QD in a 28-day treatment cycle in dose expansion component on an empty stomach or at least 1 hour after eating.
Arm/Group | Phase 1: Group 1: Lenvatinib: 12 mg | Phase 1: Group 1: Lenvatinib: 16 mg | Phase 1: Group 2: Lenvatinib: 8 mg | Phase 1: Group 2: Lenvatinib: 12 mg | Phase 2: Lenvatinib: 12 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 1/6 | 1/5 | 32/46
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/3 | 3/6 | 3/5 | 22/46
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/6 | 5/5 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Group 1: Lenvatinib: 12 mg (N=6) | Phase 1: Group 1: Lenvatinib: 16 mg (N=3) | Phase 1: Group 2: Lenvatinib: 8 mg (N=6) | Phase 1: Group 2: Lenvatinib: 12 mg (N=5) | Phase 2: Lenvatinib: 12 mg (N=46)
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 5
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Group 1: Lenvatinib: 12 mg (N=6) | Phase 1: Group 1: Lenvatinib: 16 mg (N=3) | Phase 1: Group 2: Lenvatinib: 8 mg (N=6) | Phase 1: Group 2: Lenvatinib: 12 mg (N=5) | Phase 2: Lenvatinib: 12 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 16
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1 | 13
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 10
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 3
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3 | 2 | 5
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 19
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 6 | 3 | 20
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 4 | 16
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 2 | 1 | 11
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 11
Fatigue (General disorders) | 5 | 3 | 5 | 5 | 25
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 5 | 1 | 16
Pyrexia (General disorders) | 2 | 1 | 3 | 1 | 10
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 4 | 4 | 3
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 13
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Proctitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 0 | 3 | 5
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 0 | 2 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 5 | 1 | 2 | 1 | 12
Blood urine present (Investigations) | 1 | 0 | 1 | 0 | 9
C-reactive protein increased (Investigations) | 2 | 1 | 1 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0 | 2 | 4
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 5
Thyroxine free decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Thyroxine free increased (Investigations) | 1 | 0 | 0 | 0 | 0
Tri-iodothyronine free decreased (Investigations) | 2 | 1 | 0 | 1 | 0
Tri-iodothyronine free increased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 1 | 3 | 2 | 14
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 0 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 2
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 3
Occult blood (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 8
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2 | 3 | 5 | 28
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1 | 6
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 9
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1 | 10
Proteinuria (Renal and urinary disorders) | 2 | 2 | 1 | 2 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 3 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 3 | 3 | 2 | 30
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 1 | 14
Hypertension (Vascular disorders) | 5 | 3 | 3 | 4 | 35
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2 | 2 | 11
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5
Disuse syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 3
General physical health deterioration (General disorders) | 0 | 0 | 1 | 2 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes